CLINICAL TRIAL: NCT06787729
Title: Motivation-Induced Movement Therapy: Enhancing Upper Limb Engagement in Stroke Survivors Through Ring Sensors and Data Visualization.
Brief Title: At Home Wearable Sensors and Smartphone for Stroke Survivors With Upper Limb Motor Challenges.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: University of Massachusetts, Amherst (Other); University of Maryland, College Park (Other); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Principal Investigator, Paolo Bonato, Director of Motion Analysis Laboratory, Spaulding Rehabilitation Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024P003628; 5R01EB027777-05 (NIH)
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Stroke
Keywords: Hemiparesis; Upper extremity; Weakness; Arm; Hand; Ring Sensor; Wrist Sensor; mHealth; Stroke; Activities of daily living
MeSH Terms: conditions — Stroke; Paresis; Asthenia

STUDY DESIGN:
Intervention Model Description: We will use the A (Baseline)-B (Intervention)-A (Retention) or Reversal Design. Each participant will serve as their own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mHealth Intervention (Experimental): Members of this group will receive the wearable sensors and mHealth smartphone application.
  Interventions: Device: mHealth

INTERVENTIONS:
Device: mHealth — The experimental design is composed of three phases: baseline, intervention, and retention. During the first two weeks (baseline), subjects will wear sensors, but no additional features (e.g., feedback, goal-setting, and weekly Zoom calls with clinicians) will be provided. For the next four weeks (intervention), subjects will wear sensors and have access to all intervention features, including weekly Zoom calls and goal-setting with clinicians. They will be encouraged to use the more impaired arm as much as possible. In the final two weeks (retention), the mobile intervention and clinician interactions will be removed, while subjects continue to wear sensors to examine the effects of withdrawing feedback.

SUMMARY:
The goal of this clinical trial is to learn if wearable sensor data visualization on smartphones can improve the use of the stroke-affected limb during everyday activities. Chronic stroke survivors (>12 months from onset) ages 18-80 years old with residual upper extremity motor impairments may be eligible to participate. The main question it aims to answer is:

Does the mobile health (mHealth) intervention help to improve the use of the stroke-affected upper-limb during daily living?

The study is designed so each participant serves as their own control. Researchers will compare information from the baseline, intervention, and retention time periods to see if visualizing the data on the smartphone impacts the participant's daily use of the arm.

Participants will be asked to wear a set of wearable ring and wrist sensors and interact with a custom-designed smartphone app, aiming to increase the use of their stroke-affected limb during daily activities as much as possible. They will receive feedback from the app, communicate with study therapists, participate in goal setting, complete clinical assessments, and share about their experience using the system during a virtual interview.

DETAILED DESCRIPTION:
To test the efficacy of the mHealth intervention elements (i.e., feedback, goal setting, and communication), we will use the A (Baseline)-B (Intervention)-A (Retention) or Reversal Design. The A-B-A design allows for an analysis of the effects of the introduction and subsequent removal of the intervention elements, while providing all participants an opportunity to experience the novel intervention components.

During the baseline phase (week 0 - week 2), study participants will wear the wrist and index finger-worn sensors, bilaterally, for a total of 14 days. The app will also allow study participants to self-annotate their activities approximately every 90 minutes.

During the intervention phase (week 2 - week 6), study participants will be asked to wear the wrist and/or index finger-worn sensors, bilaterally, for the next 4 weeks, similar to the baseline phase. The primary difference is that the patient will be asked to actively interact with the Intervention app, which will provide visualization of the patient's limb activity level. The platform will send auto-reminders to subjects every day at their preferred morning time to remind them to wear the wearable sensors and interact with the app. Using the sensor data collected from the wearable devices, the app will visualize the daily and weekly summary of the participants' limb activity data and the goals set by the therapist and patient. Additionally, the app will allow participants to annotate their activities and show the annotations along with the data. During the intervention phase, the participant will engage in 3 separate Zoom calls with a research therapist to 1) review the limb activity during the week, 2) discuss barriers to using the more impaired arm and ways to overcome them, 3) adjust the goal setting for the following week, and 4) document the discussions.

During the retention phase (week 6 - week 8), participants will be asked to wear the wrist and/or index finger-worn sensors, bilaterally, for the next 2 weeks. However, the mobile intervention and clinician interactions (i.e., weekly Zoom calls) will be removed, while participants continue to wear sensors to examine the effects of withdrawing feedback.

Clinical assessments will be completed after enrollment and following each phase.

ELIGIBILITY:
Inclusion Criteria:

* Stroke survivor (ischemic or hemorrhagic), >12 months post stroke, at the time of consent
* Aged between 18 and 80
* Ability to extend ≥ 10° at the metacarpophalangeal joint and one of the interphalangeal joints of each finger, ≥ 10° extension or abduction of the thumb, and ≥ 20° extension of the wrist from a fully flexed starting position.
* Demonstrating more affected arm nonuse, defined as a MAL-AoU score of < 2.5.
* Actively uses at least one smartphone app.
* Strong beliefs towards being in control of their recovery, indicated by a score of ≤ 10 points on the Internal Recovery Locus of Control (I-RLOC) Scale.
* Participants must be able to read, write, and understand English at a level sufficient to comprehend study materials and provide informed consent.

Exclusion Criteria:

* Cognitive impairments that may affect the ability to understand and follow instructions (score < 24 in the Mini Mental State Examination)
* Difficulties comprehending numbers, dyslexia, severe aphasia, or other neurological conditions that prohibit the use of smartphones for safety reasons.
* Undergoing other types of motor therapy during the study period.
* Previous participation in constraint-induced movement therapy.
* Currently participating in or has participated in the past 3 months in any experimental rehabilitation or drug studies.
* Use of botulinum toxin for motor disability ≤ 3 months before treatment.
* Significant changes in pharmacological or treatment plans during the study period that may affect upper-limb use.
* Major medical problems that could interfere with participation.
* History of a disabling stroke (i.e., need more than minimum assistance to perform ADLs).
* Legally blind status.
* Uncontrolled seizures.
* Inability to don/doff sensors independently or with the assistance of a caregiver.
* Implantable medical devices that do not comply with the ISO 14117:2012 and/or ANSI/AAMI PC69 standards for electromagnetic compatibility. Subjects will be asked to provide their medical device record card, and non-compliant devices will result in exclusion from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Motor Activity Log - Amount of Use | Week 0, Week 2, Week 6, Week 8
  This outcome measure assesses upper extremity function and use through patient report.
  Items are scored using a 6-point ordinal scale.
  For the Amount Scale, 0=the weaker arm was not used at all for that activity (not used), while 5=the weaker arm was used as often as before the stroke (same as pre-stroke).
  The score is calculated by adding the rating scores for each item and dividing by the number of items asked.
Use Duration | From enrollment to the end of the retention period at 8 weeks
  This measure evaluates the duration for which a patient actively uses their stroke-affected limb during daily activities, as recorded by a wearable accelerometer placed on the stroke-affected index finger. The unit is minutes, with a range from 0 to 3600. A value of 0 indicates no use of the stroke-affected limb during the 24-hour period, while 3600 indicates continuous activity of the limb throughout the day. To compute Use Duration, the continuous accelerometer data is segmented into short intervals (e.g., one second), and the duration is calculated by counting the time intervals where the acceleration magnitude exceeds a threshold (e.g., > 1.134 g).

SECONDARY OUTCOMES:
Motor Activity Log - Quality of Movement | Week 0, Week 2, Week 6, Week 8
  This outcome measure assesses upper extremity function and use through patient report.
  Items are scored using a 6-point ordinal scale.
  For the How Well Scale, 0=the weaker arm was not used at all for that activity (not used), while 5=the ability to use the weaker arm for that activity was as good as before the stroke (normal).
  The score is calculated by adding the rating scores for each item and dividing by the number of items asked.
Use Ratio | From enrollment to the end of the retention period at 8 weeks
  This measure compares the activity levels of the stroke-affected limb to the less-affected limb. The range is from -log(3600) to log(3600). where -log(3600) indicates exclusive use of the stroke-affected limb, log(3600) indicates exclusive use of the less-affected limb, and 0 represents equal use of both limbs. Use Ratio is computed by first determining the Use Duration for both the stroke-affected and less-affected limbs using wearable accelerometers placed on their respective index fingers. The relationship is then calculated as the logarithm of the ratio of Use Durations: log(stroke-affected use duration/less-affected use duration).

OTHER OUTCOMES:
Fugl-Meyer Assessment, Upper Extremity - Motor | Week 0, Week 2, Week 6, Week 8
  This is a motor function assessment for stroke survivors who have hemiplegia.
  Items are scored on a 3-point ordinal scale where 0=cannot perform, 1=performs partially, and 2=performs fully.
  Higher scores are indicative of higher function. Maximum score=66.
Wolf Motor Function Test - Functional Ablility | Week 0, Week 2, Week 6, Week 8
  This assessment evaluates motor ability of the upper extremity during timed and functional tasks.
  Functional ability scores are assigned using a 6-point ordinal scale, and the maximum score is 75. A score of 0=does not attempt with the involved arm and a score of 5=arm does participate; movement appears to be normal. Higher scores are indicative of higher function.
Wolf Motor Function Test - Performance Time | Week 0, Week 2, Week 6, Week 8
  This assessment evaluates motor ability of the upper extremity during timed and functional tasks.
  Performance time is measured in seconds, with up to 120 seconds allowed.
Box and Block Test | Week 0, Week 2, Week 6, Week 8
  The test is an assessment of unilateral gross manual dexterity. It is performed with each hand separately, the stroke-affected hand and the non-affected hand.
  The scored is calculated by counting the number of blocks that were carried over the partition from one side of the box to the other side of the box in 1 minute. Higher scores are indicative of better gross manual dexterity.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bonato, PhD, Principal Investigator — Director of Motion Analysis Laboratory
Locations (1):
- Spaulding Rehabilitation Hospital, Motion Analysis Laboratory, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
This is not included in the study participant consent form.